CLINICAL TRIAL: NCT05383586
Title: Inter-personal Brain Coupling Between Preterm Infants, Their Parents and a Musician During Creative Music Therapy Using Functional Near-infrared Imaging (fNIRI) Hyperscanning
Brief Title: MusicHyperBrain Study With Preterm Infants and Their Parents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-02414
Record Dates: First submitted 2022-04-19; First posted 2022-05-20 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Pre-Term
Keywords: music therapy; preterm infants; preterm parents; synchronization; hyperscanning; NIRS; HRV; oxyPrem
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: One single group will be included with a pre-during-post intervention design.
Masking Description: The intervention can not be masked since it is provided with live music to the infants and parents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Creative Music Therapy (Experimental): 20 minutes of infant-directed singing in lullaby-style accompanied with the monochord for preterm infant and parent during kangaroo-care
  Interventions: Other: Creative Music Therapy

INTERVENTIONS:
Other: Creative Music Therapy — Creative Music Therapy is provided during kangaroo-care. It is an individualized, family- centered approach offering infant-directed humming and singing accompanied with the monochord.

SUMMARY:
Inter-personal brain coupling between preterm infants, their parents and a musician during Creative Music Therapy using functional near-infrared imaging (fNIRI) hyperscanning and systemic physiology measurements

DETAILED DESCRIPTION:
Background Preterm infants represent a growing population in health care. Unfortunately, many infants suffer from neurodevelopmental impairments that persist into adolescence and adulthood. Besides other risk factors, auditory deprivation (e.g., the lack of exposure to regular intrauterine rhythms of the maternal heartbeat and the maternal voice), and the overwhelming stressful auditory environment of an intensive care unit may negatively impact brain maturation. Studies showed that infant-parent separation can impede the bidirectional development of physical, emotional, and psychological bonds between parents and their infants. Brain development is linked to nurturing social contact and early auditory experience, as demonstrated by human and animal studies. New studies showed, music is promoting neurobiological processes and neuronal learning in the human brain, which starts before birth.

Rationale Creative Music Therapy (CMT) provides meaningful interactions and a nurturing enrichment of the auditory environment by infant-directed singing in lullaby-style. Positive short-term music therapy outcomes (i.e., arousal, behavior, respiratory rate, maternal anxiety) have been shown in several reviews. Preliminary results of a recent pilot feasibility randomized controlled trial (RCT) suggest that functional brain connectivity as measured by resting-state functional magnet resonance imaging seems to have a possible early beneficial effect of CMT which manifests in (1) lower thalamo-cortical processing delay, (2) stronger functional networks, and (3) higher functional integration in predominantly left prefrontal, supplementary motor and inferior temporal brain regions. Depressive symptoms may be decreased and physical connectedness increased between infants and their parents with CMT. However, real time evaluation of CMT's possible immediate effect on the brain activity in infants and inter-personal synchronization processes between parents and infants have not been conducted yet.

The primary objective is to explore if CMT:

Improves inter-personal interaction between the infant, the parent (i.e. the mother or father) and the music therapist assessed via cerebral oxygenation synchronization between the infant and parent as well as the infant and the music therapist in the left auditory cortex and frontal cortex.

The secondary objectives are to explore if CMT:

* synchronizes inter-personal emotional/ stress responses between infant, parents (and music therapist)
* improves/ regulates brain activity in the infants' left auditory cortex and frontal cortex (evidenced by less fluctuations of cerebral hemodynamics and oxygenation)
* reduces stress in the infants
* reduces stress in the parents (mother or father)

Additionally, we aim to explore the parental perspective of CMT and their study participation.

Primary endpoint*:

Inter-personal synchronization of cerebral oxygenation and hemoglobin concentration in the brain between the infant and the parent as well as the infant and the music therapist measured by functional near-infrared spectroscopy (fNIRS) neuroimaging with a commercially available device approves for clinical applications (OxyPrem) in the left auditory and prefrontal cortex

Major secondary endpoints*:

* Inter-personal synchronization/ coupling of systemic physiology (emotional/ stress responses) in the infant and the parent as well as in the infant and the music therapist measured by systemic physiological parameters (heart rate (HR), electrodermal activity (EDA), heart rate variability (HRV), respiration rate (RR))
* Cerebral oxygenation activation/ regulation in the infant measured by fNIRS neuroimaging with OxyPrem in the left auditory and prefrontal cortex
* Stress level in the infants measured by systemic parameters (HR, EDA, HRV)
* Stress level in the parents measured by systemic parameters (EDA, HRV)
* Parental perspective of CMT and study participation

  * 15 minutes before CMT (5 minutes without kangaroo/ 10 minutes in kangaroo), 20 minutes during kangaroo with CMT, and 10 minutes after CMT (10 minutes in kangaroo/ without kangaroo)/ first session of CMT during neonatal intensive care hospitalization in the second/third week after the preterm infant's birth

Intervention:

Once/second time 20 minutes CMT: entrained infant-directed live lullaby singing, accompanied with the vibro-acoustic monochord provided by the music therapist for infant and parents in kangaroo care as described in the published clinical practice protocol.

N= 20 infant-parent couples (effect size: 1.4; significance level: 0.05; power: 0.8)

Study duration:

* Preparatory phase (months): 3 months
* First patient to last patient in/recruitment/ intervention phase: 12 months
* analysis: 2 months
* Preparation publication: 3 months Duration of the entire trial (preparatory phase + study phase): 18 months

Statistical considerations:

Brain-to-brain coupling will be determined by coherence analysis based on the fNIRS signals measured. The time-dependent coherence changes will be analyzed statistically in order to see stat. significant changes during the task compared to the baseline. Synchronization of systemic physiological signals will be determined with the same approach. Statistical analysis will be performed with ANOVA and generalized additive models (GMAs).

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable preterm infants (no invasive cardiovascular or ventilation support)
* age: 7-21 days of life
* born with 32 0/7 ≤ 36 6/7 weeks of gestation
* mentally stable parents of the included infants

Exclusion Criteria:

* admission for palliative care
* congenital malformation
* parental psychiatric disorders
* parental language barriers

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Inter-personal synchronization of cerebral oxygenation and hemoglobin concentration | 50 minutes
  Inter-personal synchronization (determined by the time-dependent coherence calculated via Wavelet transform coherence) of cerebral oxygenation (StO2 in %) and total hemoglobin concentration ([tHb] in relative µM) time-series in the brain between the infant and the parent as well as the infant and the music therapist measured by functional near-infrared spectroscopy (fNIRS) neuroimaging with a commercially available device approves for clinical applications (OxyPrem) in the left auditory and prefrontal cortex. Both devices provide similar measurements of cerebral oxygenation and hemodynamics, i.e. relative changes in the concentration of oxyhemoglobin ([O2Hb] in relative µM) and deoxyhemoglobin ([HHb] in relative µM). These time-series will be first pre-processed (removal of artifacts, band-pass filtered (0.01-0.5 Hz)) and then analyzed (Wavelet coherence and subsequent statistical analysis via a generalized additive model and Bayesian analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Bassler, Prof., Study Director — University Hospital Zurich, Department Neonatology
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No